CLINICAL TRIAL: NCT06004726
Title: "Effectiveness of School-based Substance Abuse Prevention Programme (SSPP) on Awareness, Attitude, Peer Pressure, and Life Skills Among Adolescents in Selected Public Schools of Pokhara, Nepal-A Cluster Randomized Trial"
Brief Title: "Effectiveness of School-based Substance Abuse Prevention Programme Among Adolescents .
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manipal College of Nursing (Other)
Collaborators: Manipal University (Other)
Responsible Party: Principal Investigator, Sandhya Shrestha, Principal investigator (phD Scholar), Manipal College of Nursing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 220500003
Record Dates: First submitted 2023-08-13; First posted 2023-08-22 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental and control (Experimental): Experimental group will get 4 module of intervention
  Interventions: Other: School-based Substance abuse Prevention Programme (SSPP)
- Control (No Intervention): control group will not get intervention ,Information Booklet and video assisted teaching will be given after posttest

INTERVENTIONS:
Other: School-based Substance abuse Prevention Programme (SSPP) — Module 1 :Introduction
  * Orientation about Training Programme using PowerPoint slides
  * Psychoeducation and Video Assisted Teaching to enhance awareness of substance abuse.
  * Distribution of informational booklet on basics about substance abuse
  Module 2:
  * Role play to develop a positive attitude towards the prevention of substance abuse.
  * Case-based scenario to increase resistance to peer pressure.
  * Demonstration of drug refusal techniques.
  Module3:• Storytelling on Life skills Training Components (Problem solving, Emotion Management)
  Module 4:• Demonstration of Life skills training components (Communication skills, Decision making skills, Creative thinking skills, Stress Management strategies )
  Arms: Experimental and control

SUMMARY:
The objectives of the study is to

1. "to explore the perception of teachers, parents & students in the prevention of substance abuse among adolescents".
2. "to develop and determine the effectiveness of a School-based substance abuse Prevention Programme (SSPP) on awareness, attitude, peer pressure, and life skills towards prevention of substance abuse".

In this study, SSPP refers to a Bilingual Multicomponent Training Programme which includes psychoeducation and video-assisted teaching to enhance awareness of substance abuse, role-play to develop a positive attitude towards prevention of substance abuse, Case based scenario to increase resistance to peer pressure and storytelling and demonstration to increase life skills towards prevention of substance abuse among adolescents of selected schools of Pokhara, Nepal.

DETAILED DESCRIPTION:
DETAILED METHODOLOGY

Phase I:

* Research Design: Qualitative
* Research Setting: Selected public schools of Pokhara, Nepal
* Population: Teachers, Parents, and Students of Pokhara, Nepal
* Samples: Selected Teachers, Parents & students
* Sample Size: 38 (The sample will be collected till data Saturation)
* Data collection Technique: Focus group discussion
* Data collection Tool: Focus group lead questions
* Data Analysis: Thematic analysis (Atlas.ti) Phase II Research design: Cluster Randomized Trial Randomization method: Cluster Randomization Research Setting: Selected public schools of Pokhara, Nepal Population: Adolescent students of Pokhara, Nepal Sample: Selected Adolescents, who are in the age group 13-15 years old and studying in 8th & 9th grades Variables
* Independent variables: School-based Substance abuse Prevention Programme (SSPP)
* Dependent variables: awareness, attitudes, peer pressure, and life skills related to prevention of substance abuse.
* Demographic variables: age in years, gender, religion, education/grade, family type, residence, number of siblings, education of parents, occupation of parents, sources of information, history of substance abuse in the family.

Sample size: 210

The expected outcomes of the study is to enhance awareness towards prevention of substance abuse,develop a positive attitude towards the prevention of substance abuse,develop drug refusal skills among adolescents,improve life skills and helps in th reduction of drug abuse behaviour adolescents

ELIGIBILITY:
Inclusion Criteria:

* Adolescents of 13-15 years age group.
* Those who are studying in selected public Schools of Pokhara, Nepal.

Exclusion Criteria:

* o Adolescents who are not willing to provide informed consent (assent) and parental consent.

  * Adolescents who do not belong to Nepal.
  * Adolescents who are absent during data collection

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline awareness towards substance abuse | Baseline,3months &6mobths
  Awareness towards substance abuse among adolescents using structured awareness towards substance abuse using structured awareness towards substance abuse which is of 30 items multiple choice questions with one right answer & three distracters. Higher the score higher awareness towards substance abuse
Change from baseline attitude at 3 & 6 months | Baseline,3months & 6months
  Attitude towards substance abuse using Alcohol & drug attitude scale which is of 28 items.minimum score is 61 ,Higher score is 86.higher scores indicate higher attitude t towards using Alcohol and drug
Change from baseline peer pressure at 3months & 6months | Baseline,3months& 6months
  Peer pressure towards substance abuse using peer pressure scale which is of 25 items scale.the minimum score is 55 & higher score is more than 72.higher the score high peer pressure.
Change from baseline lifeskills at 3months and 6months | Baseline,3months & 6months
  Life skills among adolescents using life skills evaluation questionnaire .Higher score indicates higher life skills.

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Shrestha, Principal Investigator — Manipal
Locations (3):
- Nepal (3):
  - Sandhya Shrestha, Pokhara, Gandaki
  - Bal mandir Mavi and Bindobasini Ma vi, Pokhara, Gandaki
  - Sandhya shrestha, Pokhara, Gandaki

IPD SHARING:
Plan to Share IPD: No